CLINICAL TRIAL: NCT04395794
Title: SARS-CoV-2 Positive Carriers Among Asymptomatic meDIcal employeeS in hiGh-volUme cardIovaScular cEnter
Brief Title: SARS-CoV-2 Disguise Study
Acronym: Disguise
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: CS-COVID-19
Record Dates: First submitted 2020-05-19; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — COVID-19 Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medical Employees: Asymptomatic medical employees in high-volume cardiovascular center.
  Interventions: Diagnostic Test: SARS-CoV-2-test; Other: SARS-CoV-2 questionnaire survey

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2-test — Nasopharyngeal and oropharyngeal testing for SARS-CoV-2
Other: SARS-CoV-2 questionnaire survey — Questionnaire regarding SARS-CoV-2 symptoms and contact with COVID patients

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection is a pandemic disease with worldwide spreading. Limited data are existed regarding SARS-CoV-2 positive carriers among asymptomatic medical employees in non-profile infectious clinic, e.g. cardiovascular clinic, routinely working in the pandemic region with two million inhabitants. The aim is to test the percentage and increase of the SARS-CoV-2 positive carriers among asymptomatic medical employees in high-volume cardiovascular center in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic medical employees of E. Meshalkin National Medical Research Center of the Ministry of Health of the Russian Federation
* Filled questionnaire before SARS-CoV-2 testing
* Nasopharyngeal and oropharyngeal testing for SARS-CoV-2
* Signed informed consent

Exclusion Criteria:

* Unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asymptomatic medical employees in high-volume cardiovascular center
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-05-07 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 positive test | 8 weeks
  Percentage of SARS-CoV-2 positive tests and increase of SARS-CoV-2 positive test between 1 st , 2 nd and 3 rd time frame testing

SECONDARY OUTCOMES:
Transformation | 8 weeks
  Percentage of transformation from asymptomatic SARS-CoV-2 positive carriers to symptomatic form
Predictors (asymptomatic) | 8 weeks
  Predictors of the asymptomatic SARS-CoV-2 positive carriers
Predictors (symptomatic) | 8 weeks
  Predictors of symptomatic form transformation
Percentage from different departments | 8 weeks
  Percentage of employees from different departments with SARS-CoV-2 positive carriers

CONTACTS AND LOCATIONS:
Locations (1):
- Meshalkin National Medical Research Center, Novosibirsk, Russia